CLINICAL TRIAL: NCT02778048
Title: Assessment of Anatomic, Physiologic and Biomechanical Characteristics of the Anal Canal and Pelvic Floor - An Observational Single Center Study on Patients Suffering From Fecal Incontinence.
Brief Title: BAFIARS - Biomedical Assessment of Function and Imaging of the Ano-rectal Sphincter
Status: Suspended | Type: Observational
Why Stopped: Funding problems
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Nano-Tera.ch, Lausanne (Unknown); Kantonsspital Winterthur KSW (Other); University of Bern (Other); University of Basel (Other)
Responsible Party: Sponsor
Other Study IDs: KEK BE 359/15
Record Dates: First submitted 2016-04-29; First posted 2016-05-19 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence | interventions — Magnetic Resonance Spectroscopy; CASP8 and FADD-Like Apoptosis Regulating Protein

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- fecal incontinence patients (m/f): patients suffering from fecal incontinence (m/f) are going to be assessed via MRI, US, FLIP, and HRAM
  Interventions: Other: MRI (magnetic resonance imaging); Other: US (ultra sound); Other: FLIP (functional lumen imaging probe); Other: HRAM (high resolution anal manometry)

INTERVENTIONS:
Other: MRI (magnetic resonance imaging) — Assessment of the sphincter
Other: US (ultra sound) — Assessment of the sphincter
Other: FLIP (functional lumen imaging probe) — Assessment of the sphincter
Other: HRAM (high resolution anal manometry) — Assessment of the sphincter

SUMMARY:
With the project Smart Muscle for Incontinence Treatment (SMIT) a multidisciplinary consortium consisting of representatives ranging from clinical medicine via microelectronics towards biomaterial science aims to develop a novel implant to treat faecal incontinence. The aim of this campaign includes development of implantable prototype devices acting as artificial continence muscles using low-voltage electrically activated polymers (EAPs) controlled by implemented pressure sensors and the patient.

Subsequently, the knowledge of the anatomical and biomechanical properties of the anal sphincter complex are of cardinal importance. Most of the existing data on anatomy and physiology results is based on old studies and almost no data on biomechanical properties are available. However, new technologies or even merging data from different examination methods might provide new information in this field.

DETAILED DESCRIPTION:
Background Fecal incontinence (FI) is affecting self-confidence and can lead to social isolation and even loss of employment Often conservative treatment as the first option is ineffective and surgical interventions follow conservative are necessary. Small defects of the anal sphincter muscles might be treated with sphincter repair and sacral neuromodulation (SNM) However, patients rarely become fully continent or short-term results deteriorate in the long term. Those patients and patients with large defects are candidates for a neosphincter procedure (artificial bowel sphincter or graciloplasty). However, the success rate of these methods is limited and the explantation rate is high. A permanent colostomy associated with massive psychosocial impairment remains as ultimate treatment option With the project Smart Muscle for Incontinence Treatment (SMIT) a multidisciplinary consortium consisting of representatives ranging from clinical medicine via microelectronics towards biomaterial science aims to develop a novel implant to treat faecal incontinence. The aim of this campaign includes development of implantable prototype devices acting as artificial continence muscles using low-voltage electrically activated polymers (EAPs) controlled by implemented pressure sensors and the patient. Subsequently, the knowledge of the anatomical and biomechanical properties of the anal sphincter complex are of cardinal importance. Most of the existing data on anatomy and physiology results is based on old studies and almost no data on biomechanical properties are available. However, new technologies or even merging data from different examination methods might provide new information in this field. Accurate imaging data on the pelvic floor region is crucial for the development of a new, implantable device for restoration of fecal continence. Optimal size (inner, outer diameter, length) and geometrical shape (cylinder, cone, torus) adapted to different functional states (rest, squeezing, defecation) will improve function and prevent erosion and consequent infection of such a prosthesis. With this study, the investigators aim to correlate three-dimensional endoanal ultrasonographic images with MRI images. The combination of different imaging techniques has been demonstrated to eliminate individual drawbacks of the examination methods and therefore would allow a precise description of the tissue. The registered data with their complementary information would permit the distinct segmentation and three-dimensional presentations of the anatomical structures in the pelvic area. This information has a great potential to facilitate diagnostics and surgical planning in this region. High-resolution anal manometry (HRAM) provides intra-anal pressure during rest or maximum pressure with high spatial and time resolution. However Biomechanical properties of the anal canal as elasticity or stiffness (compliance or flexibility) of the tissue representing important parameters for a continence organ are not routinely evaluated in daily clinical practice. Functional Lumen Imaging Probe (FLIP) allows the measurement of a cross sectional area (CSA) with respect to applied luminal pressure, respectively. FLIP has the potential to be useful in order to assess the biomechanical properties of the sphincter region. Such information potentially gives new insights in physiology and pathophysiology of the continence process. With this pilot study, the investigators aim to acquire anatomical and biomechanical data using established (manometry) and novel technologies (merging endoanal ultrasound and MRI data) in 50 patients suffering from Fecal Incontinence.

Objective Primary objective is to collect anatomical, physiological and biomechanical characteristics of the continence organ (sphincters and pelvic floor) in patients suffering from fecal incontinence and to compare this data with data gathered in an earlier study (NCT02263170) on healthy volunteers.

Secondary objectives are: test feasibility of FLIP in measuring the biomechanical properties of the anal canal and test feasibility of merging 3D US data and MR images.

Methods For the assessment of the morphology ultra sound and MRI will be used, whereas FLIP (functional luminance imaging probe) and HRAM (high resolution anal manometry) are the modality of choice to investigate the biomechanical properties of the sphincter complex.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Wexner score >= 12
* Longo's obstructed defecation syndrome (ODS) score =0
* MRI safety (no metallic implants. Appendix MRI safety form)
* Normal weighted (20<BMI<30)
* Age ≥ 60 years

Exclusion Criteria:

* Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.)
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited by flyers and advertisement in internet.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
sphincter closing pressure [mmHG] | 1 year
  at rest and during squeeze manoeuvres
sphincter muscle length [mm] | 1 year
sphincter muscle thickness [mm] | 1 year
sphincter compliance [mm/mmHG] | 1 year
  The compliance is a measure used in medicine describing the elasticity of tissue. In the case of this study it describes the elasticity of the anal canal, the sphincter muscles respectively. The compliance is directly measured with the help of the functional lumen imaging probe (FLIP).

SECONDARY OUTCOMES:
Young's modulus of sphincter muscle (mmHG/mm2] | 1 year
  combination of compliance and anatomical properties

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Brügger, PD, Dr. med., Principal Investigator — University of Bern
Locations (1):
- University Hospital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No